CLINICAL TRIAL: NCT06126133
Title: Near Infrared Spectroscopy (NIRS) Evaluation of Lumbar Plexus Block Success for Lower Extremity Orthopedic Surgery
Brief Title: Evaluation of Lumbar Plexus Block Success With Near Infrared Spectroscopy (NIRS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-6/5
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Nerve Block; Lumbar Plexus; Near Infrared Spectroscopy
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Near İnfrared Spektroskopi (NIRS) (Experimental): Peripheral oxygen saturation to be measured with NIRS device
  Interventions: Device: Near Infrared Spectroscopy

INTERVENTIONS:
Device: Near Infrared Spectroscopy — Two NIRS probes will be attached to the extremity to be operated on and to the other lower extremity on the opposite side, at a level approximately coinciding with the midline above the quandriceps femoris muscle.

SUMMARY:
Tests such as the pin-prick test, cold application or the Bromage scale are currently used to measure the success of nerve blocks and are considered subjective assessments as they require verbal consent from the patient.

Near Infrared Spectroscopy (NIRS) measures the differential absorption and reflection of near infrared light transmitted by human tissues, providing a tissue-oxygen saturation index. Modern NIRS-based instruments use multiple detectors to filter spectroscopy data from skin structures to detect subcutaneous tissue oxygenation.

Successful regional anesthesia results in decreased sympathetic activity within the distribution of blocked nerves. Regional oxygen saturation (rSO2) has been shown to increase in innervated areas after sympathetic block.

DETAILED DESCRIPTION:
The aim of this study was to show whether the success of lumbar plexus block applied in lower extremity orthopedic surgeries can be evaluated by Near Infrared Spectroscopy (NIRS), which is used to measure tissue oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old
* femoral neck fracture,
* femoral shaft fracture,
* hip replacement surgery
* who will undergo velumbar plexus block will be included in the study.

Exclusion Criteria:

* BMI>40 kg/m2
* infection in the block area
* peripheral neuropathy,
* hemoglobinopathy
* peripheral vascular disease
* allergy to local anesthetics
* patients with contraindications for lumbar plexus block

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-11 (Estimated); Primary Completion 2023-12-25 (Estimated); Study Completion 2024-01-13 (Estimated)

PRIMARY OUTCOMES:
rso2 | 40 minutes
  The regional oxymetry probe will be placed in the the quandriceps femoris muscle, one on the extremity to be operated on and the other on the opposite lower extremity.

SECONDARY OUTCOMES:
sensory block level | 40 minutes
  The sensory block level will be realised by cold testing at 10 minute intervals after applying the block.
blood pressure values | 40 minutes
  systolic, diastolic and mean blood pressure values will be recorded non-invasively in mmhg.
so2 | 40 minutes
  fingertip SO2 measured by pulse oximetry

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Assoc. PhD., Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital